CLINICAL TRIAL: NCT03413891
Title: Tranexamic Acid To Reduce Bleeding in Patients Treated With New Oral Anticoagulants Undergoing Dental Extraction
Acronym: EXTRACT-NOAC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Advice from DSMB
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Peter Verhamme, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S60131
Record Dates: First submitted 2018-01-18; First posted 2018-01-29 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-02

CONDITIONS: Tooth Extraction
Keywords: Anticoagulants; Tranexamic Acid
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): 10mL water as mouthwash with white cherry flavor in oral syringes. Once before tooth extraction and 3 times daily during 3 days post-extraction (starting day after extraction).
  Interventions: Other: Placebo
- Tranexamic Acid Group (Experimental): 10mL tranexamic acid mouthwash 10% in oral syringes. Once before tooth extraction and 3 times daily during 3 days post-extraction (starting day after extraction).
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Mouthwash
  Other Names: Exacyl
  Arms: Tranexamic Acid Group
Other: Placebo — Mouthwash
  Arms: Control Group

SUMMARY:
In patients treated with direct oral anticoagulants, bleeding events during or after tooth extraction can lead to unscheduled interruption of the antithrombotic treatment and a potential increased risk of thrombo-embolic events. Therefore, an optimal strategy to minimize bleeding events after tooth extractions is required. In this study, the investigators want to assess whether adding tranexamic acid mouthwash reduces the number of bleeding events in patients treated with direct oral anticoagulants and undergoing a tooth extraction.

DETAILED DESCRIPTION:
Interventional phase IV, randomized, double-blind, placebo-controlled trial:

* Feasibility: a 3-day regimen of tranexamic acid mouthwash in patients treated with direct oral anticoagulants
* Efficacy: reduction of bleeding events after tooth extraction compared to placebo
* Safety: any non-oral bleeding or thrombo-embolic events

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for dental extraction and treated with edoxaban, apixaban, rivaroxaban or dabigatran
* Not having taken the direct oral anticoagulant on the day of the extraction
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Subjects with any condition that as judged by the Investigator would place the subject at increased risk of harm if he/she participated in the study.
* Pregnancy or lactation
* Known allergic reaction to tranexamic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verhamme, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ockerman A, Miclotte I, Vanhaverbeke M, Vanassche T, Belmans A, Vanhove J, Meyns J, Nadjmi N, Van Hemelen G, Winderickx P, Jacobs R, Politis C, Verhamme P. Tranexamic acid and bleeding in patients treated with non-vitamin K oral anticoagulants undergoing dental extraction: The EXTRACT-NOAC randomized clinical trial. PLoS Med. 2021 May 3;18(5):e1003601. doi: 10.1371/journal.pmed.1003601. eCollection 2021 May. PMID 33939696
- See also: Pmed publication — https://doi.org/10.1371/journal.pmed.1003601

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: 10mL water as mouthwash with white cherry flavor in oral syringes. Once before tooth extraction and 3 times daily during 3 days post-extraction (starting day after extraction).
  Placebo: Mouthwash
Period: Overall Study
Arm/Group | Tranexamic Acid Group | Placebo Group
Started | 108 | 114
Completed | 106 | 112
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients except those who were lost to follow-up or who had a protocol violation were included in the full analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Group | Placebo Group | Total
Number analyzed (Participants) | 106 | 112 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (8.8) | 72.7 (10.7) | 73.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 48 | 73
  Male | 81 | 64 | 145
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 106 | 112 | 218
New oral anticoagulants (NOAC) [Count of Participants; unit: Participants]
  rivaroxaban | 38 | 40 | 78
  apixaban | 29 | 33 | 62
  edoxaban | 21 | 19 | 40
  dabigatran | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants of Oral Bleeding
Description: Any oral bleeding (early or delayed; minor, clinically relevant or major)
Time Frame: 7 days: from randomization till end of follow-up
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or had a protocol deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
Participants | 28 | 32
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p = 0.72, Chi-squared; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.60 to 1.42]

2. Secondary Outcome: Procedural Bleeding Score
Description: The Procedural bleeding score assigned by operator (VAS 0-10): Visual analogue score: ranging from 0 (no bleeding) to 10 (unstoppable bleeding)
Time Frame: Day of extraction
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
score on a scale | 4 (1.78) | 4 (1.82)

3. Secondary Outcome: Early Bleeding
Description: Any oral bleeding occurring after the extraction up to and including day 1 after the extraction
Time Frame: 2 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Number; unit: bleeding events
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
bleeding events | 35 | 49
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p = 0.36, negative-binomial regression; Rate Ratio = 0.76, 95% CI 2-sided [0.42 to 1.37]

4. Secondary Outcome: Delayed Bleeding
Description: Any oral bleeding occurring between day 2 and day 7
Time Frame: 6 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Number; unit: bleeding events
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
bleeding events | 11 | 36
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p = 0.03, negative-binomial regression; Rate Ratio = 0.32, 95% CI 2-sided [0.12 to 0.89]

5. Secondary Outcome: Minor Bleeding
Description: Any oral bleeding not requiring unplanned medical contact
Time Frame: 7 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Number; unit: bleeding events
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
bleeding events | 41 | 72
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p = 0.11, negative-binomial regression; Rate Ratio = 0.60, 95% CI 2-sided [0.32 to 1.12]

6. Secondary Outcome: Clinically-relevant Bleeding
Description: Any oral bleeding requiring unplanned medical contact
Time Frame: 7 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Number; unit: bleeding events
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
bleeding events | 5 | 13
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p = 0.15, negative-binomial regression; Rate Ratio = 0.42, 95% CI 2-sided [0.13 to 1.38]

7. Secondary Outcome: Major Bleeding
Description: Any oral bleeding requiring blood transfusion, hospitalization or resulting in death
Time Frame: 7 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Number; unit: bleeding events
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
bleeding events | 0 | 1

8. Secondary Outcome: The Number of Reinterventions
Description: Any procedure in the oral cavity for the treatment of bleeding, performed by any dentist or maxillofacial surgeon
Time Frame: 7 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Number; unit: number of reinterventions
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
number of reinterventions | 7 | 13
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p = 0.37, negative-binomial regression; Rate Ratio = 0.57, 95% CI 2-sided [0.17 to 1.91]

9. Secondary Outcome: The Number of Participants With Unplanned Interruptions of Direct Oral Anticoagulant Therapy
Description: The number of particpants with unplanned interruptions of direct oral anticoagulant therapy
Time Frame: 7 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
Participants | 6 | 9
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p = 0.66, Chi-squared; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.26 to 1.91]

10. Secondary Outcome: Number of Unplanned Medical Contacts
Description: Unplanned medical contact by phone, new consultation or hospitalization with any health care professional (dentist, general practioner, maxillofacial surgeon)
Time Frame: 7 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Number; unit: number of unplanned medical contacts
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
number of unplanned medical contacts | 10 | 27
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p = 0.04, negative-binomial regression; Rate Ratio = 0.40, 95% CI 2-sided [0.16 to 0.98]

11. Other Pre Specified Outcome: Safety Outcome: Any Non-oral Bleeding
Description: Any non-oral bleeding
Time Frame: 7 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Number; unit: bleeding events
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
bleeding events | 12 | 30
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Placebo Group; Test type: Superiority; p < 0.01, negative-binomial regression; Rate Ratio = 0.37, 95% CI 2-sided [0.18 to 0.78]

12. Other Pre Specified Outcome: Safety Outcome Number of Participants With Thrombotic Event
Description: Number of participants with thrombotic events including myocardial infarction, stroke, systemic embolism and venous thrombo-embolism
Time Frame: 7 days
Population: Full analysis set: all randomized patients except for those who were lost to follow-up or who had a protocol violation.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 106 | 112
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From inclusion in the study until patients last visit:in total 7 days
Arm/Group | Tranexamic Acid Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/114
Other Adverse Events (participants affected / at risk) | 0/108 | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03413891/Prot_SAP_000.pdf